CLINICAL TRIAL: NCT02271464
Title: Phase II Randomized Study of Maintenance Treatment With Bevacizumab or Bevacizumab Plus Metronomic Chemotherapy After First-line Induction FOLFOXIRI Plus Bevacizumab for Metastatic Colorectal Cancer Patients
Brief Title: Maintenance Bevacizumab Only or Bevacizumab Plus Metronomic Chemotherapy in Advanced Colorectal Cancer
Acronym: MOMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Alfredo Falcone, Prof., Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOMA261111; 2011-006332-23 (EudraCT Number)
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer; Ist line therapy; metronimic therapy; bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintenance:BEVACIZUMAB (Experimental): Induction: FOLFOXIRI; Manteinance: Bevacizumab
  Interventions: Drug: Maintenance:BEVACIZUMAB
- Maintenance:BEVACIZUMAB+CAPECITABINE+CYCLOPHOSPHAMIDE (Experimental): Induction: FOLFOXIRI; Maintenance:BEVACIZUMAB+CAPECITABINE+CYCLOPHOSPHAMIDE(Metronomic Chemotherapy)
  Interventions: Drug: Maintenance:BEVACIZUMAB+CAPECITABINE+CYCLOPHOSPHAMIDE

INTERVENTIONS:
Drug: Maintenance:BEVACIZUMAB — Patients will be randomly assigned to receive induction chemotherapy with the G.O.N.O. FOLFOXIRI regimen plus bevacizumab:
  * BEVACIZUMAB 5 mg/kg over 30 minutes, day 1
  * IRINOTECAN 165 mg/sqm IV over 1-h, day 1
  * OXALIPLATIN 85 mg/sqm IV over 2-h, day 1
  * L-LEUCOVORIN 200 mg/sqm IV over 2-h, day 1
  * 5-FLUOROURACIL 3200 mg/sqm IV 48-h continuous infusion, starting on day 1
  with cycles repeated every 2 weeks for 4 months (8 cycles), followed after 2 weeks by (if no progression occurs):
  - BEVACIZUMAB 7.5 mg/kg over 30 minutes, day 1 (every three weeks)
  Arms: Maintenance:BEVACIZUMAB
Drug: Maintenance:BEVACIZUMAB+CAPECITABINE+CYCLOPHOSPHAMIDE — Patients will be randomly assigned to receive induction chemotherapy with the G.O.N.O. FOLFOXIRI regimen plus bevacizumab:
  * BEVACIZUMAB 5 mg/kg over 30 minutes, day 1
  * IRINOTECAN 165 mg/sqm IV over 1-h, day 1
  * OXALIPLATIN 85 mg/sqm IV over 2-h, day 1
  * L-LEUCOVORIN 200 mg/sqm IV over 2-h, day 1
  * 5-FLUOROURACIL 3200 mg/sqm IV 48-h continuous infusion, starting on day 1
  with cycles repeated every 2 weeks for 4 months (8 cycles), followed after 2 weeks by (if no progression occurs):
  * BEVACIZUMAB 7.5 mg/kg over 30 minutes, day 1 (every three weeks),
  * CAPECITABINE 500 mg/tid orally, continuously,
  * CYCLOPHOSPHAMIDE 50 mg/day orally, continuously.
  Arms: Maintenance:BEVACIZUMAB+CAPECITABINE+CYCLOPHOSPHAMIDE

SUMMARY:
This study consist of 4-months induction first-line chemotherapy with the G.O.N.O. FOLFOXIRI regimen plus bevacizumab followed by maintenance with bevacizumab or bevacizumab plus metronomic chemotherapy (with capecitabine and cyclophosphamide) in mCRC patients.

The main objective of this study is to preliminarily evaluate the potential effects of the combination of a metronomic chemotherapy with capecitabine and cyclophosphamide to maintenance bevacizumab on pharmacodynamic and clinical parameters among mCRC patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of colorectal cancer.
* Not resectable metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease.
* At least one measurable lesion according to RECIST criteria.
* Male or female of 18-75 years of age.
* ECOG PS < 2 if aged < 71 years, ECOG PS = 0 if aged 71-75 years;
* Life expectancy of at least 12 weeks.
* Previous adjuvant chemotherapy containing oxaliplatin is allowed if more than 12 months have elapsed between the end of adjuvant therapy and first relapse;
* Previous adjuvant chemotherapy with fluoropyrimidine monotherapy is allowed if more than 6 months have elapsed between the end of adjuvant and first relapse;
* Neutrophils 1.5 x 109/L, Platelets 100 x 109/L, Hgb >9 g/dl.
* Total bilirubin 1.5 time the upper-normal limits (UNL) of the institutional normal values and ASAT (SGOT) and/or ALAT (SGPT) 2.5 x UNL, or 5 x UNL in case of liver metastases, alkaline phosphatase 2.5 x UNL, 5 x UNL in case of liver metastases.
* Creatinine clearance >50 mL/min or serum creatinine 1.5 x UNL.
* Urine dipstick of proteinuria <2+. Patients discovered to have 2+ proteinuria on dipstick urinalysis at baseline, should undergo a 24-hour urine collection and must demonstrate <1 g of protein/24 hr.
* Written informed consent to treatment and translational analyses.

Exclusion Criteria:

* Radiotherapy to any site within 4 weeks before the study.
* Previous treatment with bevacizumab
* Untreated brain metastases or spinal cord compression or primary brain tumours.
* History or evidence upon physical examination of CNS disease unless adequately treated.
* Symptomatic peripheral neuropathy > 2 grade NCIC-CTG criteria;
* Serious, non-healing wound, ulcer, or bone fracture.
* Evidence of bleeding diathesis or coagulopathy.
* Uncontrolled hypertension.
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication.
* Current or recent (within 10 days prior to study treatment start) ongoing treatment with anticoagulants for therapeutic purposes.
* Chronic, daily treatment with high-dose aspirin (>325 mg/day).
* Treatment with any investigational drug within 30 days prior to enrollment.
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal and squamous cell carcinoma or cervical cancer in situ.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study (barrier contraceptive measure or oral contraception).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2012-03; Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | up to 4 years
  PFS is defined as the time from randomization to first documentation of objective disease progression or death due to any cause, whichever occurs first.PFS will be censored on the date of the last evaluable on study tumor assessment documenting absence of progressive disease for patients who are alive,on study and progression free at the time of the analysis.Alive patients having no tumor assessments after baseline will have time to event endpoint censored on the date of randomization.Disease status will be evaluated according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Best overall response rate (ORR) | up to 4 years
  It is defined as the percentage of patients,relative to the total of enrolled subjects,achieving a complete or partial response, according to RECIST 1.1 criteria,during the induction and the maintenance phases of treatment.The determination of clinical response will be based on investigator reported measurements that will be subsequently confirmed by a central review.Responses will be evaluated every 8 weeks.Patients who do not have an on-study assessment will be included in the analysis as non responders.
Duration of response | up to 4 years
  it is defined as the time from the date when measurement criteria are met for CR or PR until first documentation of objective disease progression
Resection rate | up to 4 years
  it is defined as the percentage of patients, relative to the total of enrolled subjects, undergoing secondary R0 resection of metastases during treatment or after its completion.
  Secondary R0 surgery is defined as microscopically margin-free complete surgical removal of all residual disease, allowed by tumoral shrinkage and/or disappearance of one or more lesions.
Time to strategy failure (TSF) | up to 4 years
  it is defined as the time from the day of randomization to one of the followings:
  1. progression during FOLFOXIRI + bevacizumab or during a modified FOLFOXIRI + bevacizumab regimen; OR
  2. progression and decision to not administer FOLFOXIRI + bevacizumab or a modified FOLFOXIRI + bevacizumab regimen; OR
  3. introduction of a new agent not included in the study treatment according to randomization arm; OR
  4. death; whichever occurs first.For patients still on-treatment at the time of analysis, the time to strategy failure will be censored on the last date the patients were known to be alive.
Time to 2nd progressive disease | up to 4 years
  it is defined as the time from randomization to second documentation of objective disease progression or death due to any cause, whichever occurs first.
  Time to 2nd progressive disease will be censored on the date of the last evaluable on-study tumor assessment documenting absence of progressive disease for patients who are alive, on study and second progression-free at the time of the analysis. Alive patients having no tumor assessments after baseline will have time to event endpoint censored on the date of randomization.
Overall survival (OS) | up to 4 years
  it is defined as the time from randomization to the date of death due to any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.
Toxicity rate | up to 4 years
  it is defined as the percentage of patients, relative to the total of enrolled subjects, experiencing a specific adverse event, according to National Cancer Institute Common Toxicity Criteria (version 4.0), during the induction and the maintenance phases of treatment.
Overall toxicity rate | up to 4 years
  it is defined as the percentage of patients, relative to the total of enrolled subjects, experiencing any adverse event, according to National Cancer Institute Common Toxicity Criteria (version 4.0), during the induction and the maintenance phases of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Falcone, MD, Principal Investigator — Polo Oncologico Area Vasta Nord Ovest
Locations (20):
- Italy (20):
  - Istituto Ospedaliero Fondazione Poliambulanza Di Brescia, Brescia
  - Pres.Ospedaliero Spedali Civili Brescia, Brescia
  - Istituti Ospitalieri Di Cremona, Cremona
  - Azienda Ospedaliera S. Croce E Carle Di Cuneo, Cuneo
  - A.O. Universitaria Arcispedale S.Anna Di Ferrara, Ferrara
  - Ausl Di Frosinone -, Frosinone
  - E.O. Ospedali Galliera, Genova
  - Ospedale Per Acuti Mater Salutis Di Legnago, Legnago
  - Oncologia AUSL 2 Lucca, Lucca
  - Irccs Fondazione Centro S. Raffaele Del Monte Tabor, Milan
  - A.O. Universitaria Federico Ii Di Napoli, Napoli
  - Irccs Istituto Oncologico Veneto (Iov), Padua
  - Polo Oncologico Area Vasta Nord Ovest, Pisa
  - Ausl 5 Di Pisa, Pontedera
  - Ospedale Mesericordia E Dolce, Prato
  - Ospedale S. Maria Nuova, Reggio Emilia
  - Ospedale San Giovanni Calibita Fatebenefratelli, Roma
  - Ospedale San Pietro Fatebenefratelli Di Roma, Roma
  - Campus Biomedico, Roma
  - A.O. Universitaria S. Maria Della Misericordia, Udine

REFERENCES:
- [Derived] Cremolini C, Marmorino F, Bergamo F, Aprile G, Salvatore L, Masi G, Dell'Aquila E, Antoniotti C, Murgioni S, Allegrini G, Borelli B, Gemma D, Casagrande M, Granetto C, Delfanti S, Di Donato S, Schirripa M, Sensi E, Tonini G, Lonardi S, Fontanini G, Boni L, Falcone A. Phase II randomised study of maintenance treatment with bevacizumab or bevacizumab plus metronomic chemotherapy after first-line induction with FOLFOXIRI plus Bevacizumab for metastatic colorectal cancer patients: the MOMA trial. Eur J Cancer. 2019 Mar;109:175-182. doi: 10.1016/j.ejca.2018.12.028. Epub 2019 Feb 5. PMID 30735919
- [Derived] van Dijk E, Biesma HD, Cordes M, Smeets D, Neerincx M, Das S, Eijk PP, Murphy V, Barat A, Bacon O, Prehn JHM, Betge J, Gaiser T, Fender B, Meijer GA, McNamara DA, Klinger R, Koopman M, Ebert MPA, Kay EW, Hennessey BT, Verheul HMW, Gallagher WM, O'Connor DP, Punt CJA, Loupakis F, Lambrechts D, Byrne AT, van Grieken NCT, Ylstra B. Loss of Chromosome 18q11.2-q12.1 Is Predictive for Survival in Patients With Metastatic Colorectal Cancer Treated With Bevacizumab. J Clin Oncol. 2018 Jul 10;36(20):2052-2060. doi: 10.1200/JCO.2017.77.1782. Epub 2018 May 24. PMID 29792754
- [Derived] Cremolini C, Casagrande M, Loupakis F, Aprile G, Bergamo F, Masi G, Moretto R R, Pietrantonio F, Marmorino F, Zucchelli G, Tomasello G, Tonini G, Allegrini G, Granetto C, Ferrari L, Urbani L, Cillo U, Pilati P, Sensi E, Pellegrinelli A, Milione M, Fontanini G, Falcone A. Efficacy of FOLFOXIRI plus bevacizumab in liver-limited metastatic colorectal cancer: A pooled analysis of clinical studies by Gruppo Oncologico del Nord Ovest. Eur J Cancer. 2017 Mar;73:74-84. doi: 10.1016/j.ejca.2016.10.028. Epub 2016 Dec 13. PMID 27986363